CLINICAL TRIAL: NCT07064421
Title: Non-Helium Magnetoencephalography for Clinical Management of Refractory Epilepsy in Children: An Observational Cohort Study
Brief Title: Non-Helium Magnetoencephalography in Pediatric Refractory Epilepsy
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Collaborators: Beijing X-Magtech Technology Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: 446A01
Record Dates: First submitted 2025-02-26; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Refractory Epilepsy in Children
Keywords: Epilepsy; Magnetoencephalography
MeSH Terms: conditions — Epilepsy | interventions — Magnetoencephalography; Electrocorticography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Participants in the case group will undergo both MEG and SEEG/ECoG for preoperative assessment.
  Interventions: Diagnostic Test: Magnetoencephalography plus Stereo-electroencephalography/Electrocorticography
- Control: Patients in the control group will undergo only SEEG/ECoG before surgery.
  Interventions: Diagnostic Test: Stereo-electroencephalography/Electrocorticography

INTERVENTIONS:
Diagnostic Test: Magnetoencephalography plus Stereo-electroencephalography/Electrocorticography — Use Magnetoencephalography and Stereo-electroencephalography/Electrocorticography in the preoperative assessment of children with drug-resistant epilepsy, particularly in identifying the seizure focus.
  Groups: Case
Diagnostic Test: Stereo-electroencephalography/Electrocorticography — Use Stereo-electroencephalography/Electrocorticography in the preoperative assessment of children with drug-resistant epilepsy, particularly in identifying the seizure focus.
  Groups: Control

SUMMARY:
The goal of this observational study is to evaluate the effectiveness of Magnetoencephalography (MEG) in the preoperative assessment of children with refractory epilepsy, particularly in identifying the seizure focus, and to compare it with the gold standard methods of Stereo-electroencephalography (SEEG) and Electrocorticography (ECoG).

The main questions this study aims to answer are:

1. How consistent is MEG with SEEG/ECoG in locating the epileptic focus in children with refractory epilepsy?
2. What is the clinical efficacy of MEG in identifying epileptic foci?

Participants will:

1. Be divided into 2 groups: the case group and the control group. Participants in the case group will undergo both MEG and SEEG/ECoG for preoperative assessment, while patients in the control group will undergo only SEEG/ECoG before surgery.
2. Be followed up at 1, 3, 6, and 12 months after surgery to assess seizure control, neurological function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 3-18 years old;
2. Clinically diagnosed with refractory epilepsy;
3. Capable of cooperating with magnetoencephalography evaluation and recording.

Exclusion Criteria:

1. Patients with serious comorbidities or neurological or psychiatric disorders that affect magnetoencephalography examination.
2. Patients using drugs that affect central nervous system function;
3. Patients who are not suitable for surgical procedures;
4. Patients with progressive neurological disorders.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients of Guangzhou Women and Children's Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Agreement in Epileptogenic Zone Localization Between Magnetoencephalography (MEG) and Stereoelectroencephalography/Electrocorticography (SEEG/ECoG) (Kappa Coefficient) | From enrollment to 12 months after surgery.
  This outcome measures the agreement between preoperative MEG and SEEG/ECoG (gold standard) in localizing the epileptogenic zone. Consistency will be quantified using Cohen's Kappa coefficient (κ) with 95% confidence intervals. Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) will be calculated. Data aggregation will compare MEG-derived localization (categorized by brain regions, e.g., temporal lobe, frontal lobe) with intraoperative SEEG/ECoG findings. Statistical analysis will be performed using SPSS 27.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women and Children's medical center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No